CLINICAL TRIAL: NCT00929344
Title: Duloxetine Versus Pregabalin for Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Barbara J. Mason, PI, The Scripps Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AA014028; R37AA014028 (NIH); MERIT
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-03

CONDITIONS: Alcohol Dependence
Keywords: Alcohol; Alcohol treatment; Alcoholism; Alcohol Abuse; Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Pregabalin; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Duloxetine (Experimental)
  Interventions: Drug: Duloxetine; Behavioral: Standardized behavioral therapy
- Pregabalin (Experimental)
  Interventions: Drug: Pregabalin; Behavioral: Standardized behavioral therapy
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Behavioral: Standardized behavioral therapy

INTERVENTIONS:
Drug: Pregabalin — Two 150 mg capsules, 150 mg/am and 150 mg/pm (Total dose, 300mg/d), 12 week duration. Dose may be increased up to 600 mg/d or reduced to 150 mg/d based on subject response and tolerability.
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Duloxetine — 40 mg capsule, Once daily/am, 12 week duration, placebo capsule administered pm. Dose may be increased up to 60 mg/d or reduced to 20 mg/d based on subject response and tolerability.
  Other Names: Cymbalta
  Arms: Duloxetine
Behavioral: Standardized behavioral therapy — Standardized behavioral therapy 1 time per week for 12 week duration.
  Other Names: Manually-guided therapy
  Arms: Duloxetine
Behavioral: Standardized behavioral therapy — Standardized behavioral therapy 1 time per week for 12 week duration.
  Other Names: Manually-guided therapy
  Arms: Pregabalin
Drug: Placebo — Matched placebo capsule administered 1 capsule am and 1 capsule pm for 12 week duration.
  Arms: Placebo
Behavioral: Standardized behavioral therapy — Standardized behavioral therapy 1 time per week for 12 week duration.
  Other Names: Manually-guided therapy
  Arms: Placebo

SUMMARY:
A 12-week, double-blind, placebo-controlled parallel group study will be conducted with 150 outpatients with alcohol dependence, with random assignment to pregabalin 300 mg/d, duloxetine 40 mg/d, or placebo in conjunction with manual-guided behavioral counseling and follow-up visits 1 week and 3 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age
* Meets DSM-IV criteria for current alcohol dependence and drinking an average of ≥21 drinks weekly for males, ≥14 females,
* Seeking research-based outpatient treatment for alcohol problems
* Willing to attend 12 weekly study visits and 2 follow-up visits
* Have normal bilirubin, and ALT, AST, and GGT values no more than 3x the ULN, and no evidence of hepatic insufficiency

Exclusion Criteria:

* Active suicidal ideation
* Medical disorders that will increase potential risk or interfere with study participation
* Sexually active female subjects with childbearing potential who are pregnant, nursing or refuse to use a reliable method of birth control
* Males who refuse to use a reliable method of birth control
* Meets DSM-IV criteria for any other current major AXIS I disorder other than alcohol or nicotine dependence.
* Inability to understand and/or comply with the provisions of the protocol and consent form
* Treatment with an antidepressant medication during the two weeks, or fluoxetine during the month, prior to randomization
* Ongoing treatment with disulfiram (Antabuse), naltrexone (ReVia), acamprosate (Campral) or other medications that may affect study outcomes, e.g., anticonvulsants or other drugs that act on serotonin in the brain
* Ongoing treatment with drugs that may increase potential risk (Actos),

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Mason, Ph.D., Principal Investigator — The Scripps Research Institute
Locations (1):
- The Scripps Research Institute Pearson Center for Alcoholism and Addiction Research, La Jolla, California, United States

REFERENCES:
- See also: Study Information — http://alcoholismmarijuanatreatment.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duloxetine | Pregabalin | Placebo
Started | 50 | 50 | 50
Completed | 28 | 37 | 29
Not Completed | 22 | 13 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Pregabalin | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.86 (10.53) | 44.56 (11.55) | 43.54 (10.52) | 44.32 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 23 | 55
  Male | 31 | 37 | 27 | 95

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Drinking Quantity and Frequency Using Drinks Per Week at Week 12
Description: Standard drinks are equivalent to 14 grams of pure alcohol and number of drinks are assessed with Timeline Follow-Back (TLFB) methods. Change = (Week 12 - Baseline). More negative values indicate less use of alcohol.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: drinks/week
Arm/Group | Duloxetine | Pregabalin | Placebo
Number analyzed (Participants) | 28 | 37 | 29
drinks/week
  Drinks/week Baseline | 42.07 (17.94) | 56.67 (50.93) | 41.20 (27.39)
  Drinks/week Week 12 | 9.16 (11.90) | 7.59 (15.73) | 8.06 (11.22)
  Drinks/week Change | -32.91 (20.38) | -49.08 (44.91) | -33.15 (23.32)

2. Primary Outcome: Change From Baseline in Drinking Quantity and Frequency Using Drinking Days Per Week at Week 12
Description: Standard drinks are equivalent to 14 grams of pure alcohol and number of drinks are assessed with Timeline Follow-Back (TLFB) methods. A drinking day is a day where any alcohol is consumed. Change = (Week 12 - Baseline). More negative values indicate less use of alcohol.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: drinking days/week
Arm/Group | Duloxetine | Pregabalin | Placebo
Number analyzed (Participants) | 28 | 37 | 29
drinking days/week
  Drinking Days/Week Baseline | 5.11 (1.29) | 4.54 (1.64) | 4.87 (1.60)
  Drinking Days/Week Week 12 | 2.17 (2.59) | 1.14 (1.90) | 1.85 (2.20)
  Drinking Days/Week Change | -2.94 (2.68) | -3.40 (2.03) | -3.01 (2.20)

3. Primary Outcome: Change From Baseline in Drinking Quantity and Frequency Using Drinks Per Drinking Day at Week 12
Description: as for outcome 2
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: drinks/drinking day
Arm/Group | Duloxetine | Pregabalin | Placebo
Number analyzed (Participants) | 28 | 37 | 29
drinks/drinking day
  Drinks/Drinking Day Baseline | 8.16 (2.69) | 12.98 (11.14) | 8.91 (5.41)
  Drinks/Drinking Day Week 12 | 2.21 (2.65) | 2.31 (3.81) | 2.90 (3.62)
  Drinks/Drinking Day Change | -5.94 (3.54) | -10.67 (11.34) | -6.01 (4.84)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected weekly at all 14 study visits during the double blind portion of the study, an average duration of 12 weeks. Adverse event data was also collected during two additional follow up visits, at Weeks 13 and 24.
Description: Adverse events, both serious and other, were documented at all 16 study visits by the Medical Assistant on the adverse event case report form.
Arm/Group | Duloxetine | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/50 | 0/50 | 4/50
Other Adverse Events (participants affected / at risk) | 43/50 | 35/50 | 33/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duloxetine (N=50) | Pregabalin (N=50) | Placebo (N=50)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Gastrointestinal protozoal infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Duloxetine (N=50) | Pregabalin (N=50) | Placebo (N=50)
Vision blurred (Eye disorders) | 0 | 4 | 1
Constipation (Gastrointestinal disorders) | 6 | 7 | 3
Diarrhoea (Gastrointestinal disorders) | 9 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 7 | 9 | 3
Dyspepsia (Gastrointestinal disorders) | 6 | 1 | 1
Nausea (Gastrointestinal disorders) | 9 | 6 | 2
Toothache (Gastrointestinal disorders) | 1 | 3 | 3
Fatigue (General disorders) | 2 | 3 | 4
Bronchitis (Infections and infestations) | 1 | 4 | 2
Influenza (Infections and infestations) | 5 | 2 | 2
Nasopharyngitis (Infections and infestations) | 15 | 9 | 16
Urinary tract infection (Infections and infestations) | 3 | 4 | 2
Hepatic enzyme increased (Investigations) | 4 | 0 | 0
Abnormal weight gain (Metabolism and nutrition disorders) | 0 | 3 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Disturbance in attention (Nervous system disorders) | 3 | 2 | 1
Dizziness (Nervous system disorders) | 5 | 7 | 0
Headache (Nervous system disorders) | 14 | 6 | 8
Somnolence (Nervous system disorders) | 6 | 12 | 4
Tremor (Nervous system disorders) | 0 | 3 | 0
Insomnia (Psychiatric disorders) | 6 | 3 | 1
Libido decreased (Psychiatric disorders) | 5 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No